CLINICAL TRIAL: NCT02143804
Title: Phase II Safety and Efficacy Study of CG0070 Oncolytic Vector Regimen in Patients With High Grade Non-Muscle Invasive Bladder Carcinoma Disease (NMIBC) Who Have Failed BCG and Refused Cystectomy
Brief Title: Safety and Efficacy of CG0070 Oncolytic Virus Regimen in Patients With High Grade Non-Muscle Invasive Bladder Cancer
Acronym: exBOND
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in trial design
Sponsor: CG Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: exBOND 2.1
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Bladder Cancer; High Grade; Non Muscle Invasive
Keywords: Oncolytic virus; GMCSF; pRb; PDL1; Immunotherapy; Adenovirus
MeSH Terms: conditions — Urinary Bladder Neoplasms; Adenoviridae Infections

ARMS (1):
- CG0070 (Experimental): oncolytic virus genetically modified to express GM-CSF
  Interventions: Biological: oncolytic adenovirus expressing GMCSF

INTERVENTIONS:
Biological: oncolytic adenovirus expressing GMCSF — Treatment once weekly by intravesical route. Use of DDM to first remove the GAG layer of the bladder and to improve virus transduction. Installation of 100 ml. of CG0070 at 10e12 viral particles for 45 minutes inside bladder.
  Other Names: CG0070; Adenovirus with GMCSF expression; DDM

SUMMARY:
This is an expanded access protocol to study the safety and efficacy of CG0070 in Cis and Cis with Ta and/or T1 disease patients who failed both BCG therapy and the BOND protocol (NCT 01438112), or in high grade Ta and T1 patients who failed BCG therapy.

DETAILED DESCRIPTION:
The plan is to study the safety and efficacy of CG0070 in high-grade NMIBC patients who failed BCG therapy. Most patients with NMIBCis (Cis, Cis with Ta and/or T1, high grade Ta or T1 with frequent or uncontrolled recurrences) who have failed BCG intravesical therapy (standard of care) usually have no other choice but to proceed to cystectomy. Cystectomy is a surgery associated with major morbidity, mortality and quality of life issues. Morbidity and long term tedious medical care will be for the rest of the patient's life span. Most patients at this stage do not show signs of disease progression into the muscle layer or of metastasis, making surgery a very difficult decision. CG0070, if successful in this trial, will serve to provide a therapeutic alternative for this patient population in need. For the present study, Cis or Cis with Ta and/or T1 patients can only be enrolled if they have failed the BOND study and are medically unfit for surgery. Furthermore, patients with high grade Ta or T1 disease who have failed both BCG and chemotherapy treatments are also prone to disease progression. Since these patients are not eligible to be enrolled in the BOND trial, the present study will serve as an alternative to access CG0070 experimental treatment.

ELIGIBILITY:
Inclusion Criteria:

* • Patients must have pathologically confirmed high grade disease (HG), as defined by the 2004 WHO classification system

  * Patients must have no evidence of muscle invasive disease
  * Patient must fall under one of the following criteria:

    1. Patients who were first enrolled in the BOND protocol but have failed to achieve a complete response or have relapsed following a complete response at 3 months after receiving control treatments
    2. OR patients who were first enrolled in the BOND protocol but have relapsed following a complete response lasting over a year after receiving CG0070 treatments
    3. OR patients who have Ta/T1 high grade, refused cystectomy and are CG0070 naïve
    4. OR patients from the exBOND protocol who experienced a tumor relapse with no disease progression after sustaining 12 months or longer complete response duration
  * For Cis patients or Cis with Ta and/or T1 only:

    1. Tumor must be considered unresectable or with residual disease.
    2. Patients must be declared as medically unfit for cystectomy.
    3. No disease progression from disease status at the beginning of the BOND trial.
  * For Ta/T1 HG Patients:

    1. They must have also received at least one prior course of BCG therapy per the recommended schedules. Patients can have either failed BCG induction therapy within a six-month period or have been successfully treated with BCG, but subsequently found to have recurrence. The standard course of intravesical BCG therapy must include at least six weekly treatments (allowable range of instillations per course is 4-9) within a six-month period
    2. They must have received 2 or more intravesical chemotherapy regimens other than BCG
    3. They must have relapsed within 6 months of their last treatment
  * 18 years of age or older
  * Radical cystectomy has been declined by the patient in a signed special section of the informed consent, whereby there is a clear explanation by the investigator to the subject that a delay of cystectomy may increase his/her chance of disease progression, the results of which may lead to serious and life threatening consequences.
  * Patients must be able to enter into the study within five weeks of their most recent diagnostic procedure, which is usually a diagnostic biopsy, a transurethral resection of bladder tumor (TURBT) procedure or other diagnostic scanning such as CT and PET procedures.
  * Histopathologically confirmed, transitional cell (urothelial) carcinoma. Urothelial tumors with mixed histology (but with <50% variant) are eligible.
  * Eastern Cooperative Oncology Group (ECOG) performance status <2.
  * Not pregnant or lactating
  * Patients with child bearing potential must agree to use adequate contraception
  * Agree to study specific informed consent and HIPAA authorization for release of personal health information
  * Adequate baseline CBC, renal and hepatic function. Parameters described as .WBC>3000 cells/mm3, ANC>1,000 cells/mm3, hemoglobin>10g/dL, and platelet count >100,000 cells/mm3

    * Adequate renal function: serum creatinine <2.0mg/dL
    * Bilirubin, AST and ALT not more than 2 x Upper Limits of Normal
    * PT/INR, PTT, and fibrinogen within institutional normal limits
    * Absolute lymphocyte count ≥ 800/μL before the first dose of CG0070

Exclusion Criteria:

* Previous systemic chemotherapy or radiation for bladder cancer. Note: Prior immunotherapy or intravesical (administered within the bladder) chemotherapy for superficial disease is acceptable

  * History of anaphylactic reaction following exposure to humanized or human therapeutic monoclonal antibodies, hypersensitivity to GM-CSF or yeast derived products, clinically meaningful allergic reactions or any known hypersensitivity or prior reaction to any of the formulation excipients in the study drugs.
  * Known infection with HIV, HBV or HCV.
  * Anticipated use of chemotherapy, radiotherapy, or other immunotherapy not specified in the study protocol while on study
  * Any underlying medical condition that, in the Investigator's opinion, will make the administration of study vector hazardous to the patient, would obscure the interpretation of adverse events, or not permit adequate surgical resection.
  * Systemic treatment on any investigational clinical trial within 28 days prior to registration.
  * Concurrent treatment with immunosuppressive or immunomodulatory agents, including any systemic steroid (exception: inhaled or topically applied steroids, and acute and chronic standard dose NSAIDs, are permitted). Use of a short course (i.e., ≤ 1 day) of a glucocorticoid is acceptable to prevent a reaction to the IV contrast used for CT scans.
  * Immunosuppressive therapy, including: cyclosporine, antithymocyte globulin, or tacrolimus within 3 months of study entry.
  * History of prior experimental cancer vaccine treatment (e.g., dendritic cell therapy, heat shock vaccine)
  * History of stage III or greater cancer, excluding urothelial cancer. Basal or squamous cell skin cancers must have been adequately treated and the subject must be disease-free at the time of registration. Subjects with a history of stage I or II cancer, must have been adequately treated and have been disease-free for ≥ 3 years at the time of registration.
  * Progressive viral or bacterial infection

    o All infections must be resolved and the patient must remain afebrile for seven days without antibiotics prior to being placed on study
  * Unwilling or unable to comply with the protocol or cooperate fully with the investigator and site personnel
  * Evidence of disease progression compared to disease status before BOND protocol for NMIBCis patients.
  * Patient have relapsed less than 1 year after or who are refractory to treatment with CG0070.
  * Cis, and Cis with Ta and/or T1 patients who are medically fit for cystectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Durable Complete Response Proportion | 15 month time point from the date of the first intravesical treatment and/or at least 12 months from the initial complete response assessment (3 months from first intravesical treatment) or any time after
  DCR

CONTACTS AND LOCATIONS:
Locations (1):
- BCG Oncology, Phoenix, Arizona, United States